CLINICAL TRIAL: NCT04602988
Title: Continuous, Non-Invasive Monitoring of Mental Status
Brief Title: Study to Assess and Monitor Brain Activity
Acronym: SAMBA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Eyal Y. Kimchi, M.D.,Ph.D., Assistant Professor, Massachusetts General Hospital
Other Study IDs: 2020P000678
Record Dates: First submitted 2020-10-18; First posted 2020-10-26 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Delirium; Encephalopathy
Keywords: EEG; Mental Status
MeSH Terms: conditions — Delirium; Brain Diseases | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients admitted to an inpatient hospital unit: Patients admitted to an inpatient hospital unit will receive EEG based monitoring of mental status
  Interventions: Device: EEG

INTERVENTIONS:
Device: EEG — EEG monitoring of brain rhythms

SUMMARY:
A mainstay in the diagnosis and care of hospitalized patients is the assessment of mental status. Changes in mental status can have broad clinical significance, and while some patients are admitted with mental status changes, nearly half of the patients who experience delirium in the hospital develop it after admission in a manner that is hard to predict on the level of individual patients. Patients with altered mental status such as delirium have worse clinical outcomes, suggesting that early monitoring of mental status can identify important clinical populations who may benefit from targeted delirium prevention and intervention. Delirium remains under-recognized in the hospital, in part due to its fluctuating nature. Typically, mental status is assessed sporadically, perhaps once a day, through intermittent and subjective clinical interactions. As such, there is a clear clinical need for objective, continuous methods to monitor mental status. Such methods could potentially improve detection of delirium, potentially even predicting it prior to clinical recognition, and therefore direct multimodal delirium prevention and intervention strategies when most effective-before delirium becomes fully manifest. In this proposal we plan on testing noninvasive, continuous monitors of mental status in the inpatient setting, primarily through the use of EEG.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to a general medical ward
* Expected stay of at least one night

Exclusion Criteria:

* patients who have any scalp incisions or head wound(s) that would prevent EEG attachment
* Non-English speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited after their admission to inpatient medical units at the participating hospital.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2020-08-10 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Delirium Severity | Daily during the time of EEG recording up to 7 days
  Inpatient Delirium as assessed by the 3D-CAM-S
EEG | Daily during the time of EEG recording up to 7 days
  Relative EEG power in the delta & theta bands

SECONDARY OUTCOMES:
Functional status | 3 months after completion of EEG recording
  Functional status as assessed by the Glasgow Outcome Score (1-5, with lower numbers less favorable outcomes and higher numbers more favorable outcomes)

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Y Kimchi, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided